CLINICAL TRIAL: NCT06177990
Title: Caregiver as Navigator: Develop Skills Online (CAN-DO) Developing Dementia Family Caregiver Mastery for Navigating Complex Health, Social Service, Legal, Financial, and Family Systems
Brief Title: Caregiver as Navigator: Develop Skills Online (CAN-DO)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Carolyn Clevenger, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006261; 1R01AG082833-01 (NIH)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Dementia
Keywords: Caregiver; Dementia
MeSH Terms: conditions — Dementia | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAN-DO Immediate program group (Experimental): Each participant will be engaged in a baseline interview. Subsequently, each will be asked to take part in follow-up interviews at points 2, 4, 6, and 8 months following the launch of their cohort.
  Interventions: Other: Caregiver as Navigator: Develop Skills Online (CAN-DO) program
- Attention Control program group (Active Comparator): Participants will receive an online course about "Healthy Living" for the first 4 months after randomization.
  After the Attention Control participants complete their 4-month interview, they will be invited to participate in the CAN-DO program.
  Interventions: Other: Caregiver as Navigator: Develop Skills Online (CAN-DO) program; Other: Healthy Living online course
- Usual care group (Active Comparator): Participants randomized to the Usual care group will not receive intervention from the study but after they complete their 4-month interview, they will be invited to participate in the CAN-DO program.
  Interventions: Other: Caregiver as Navigator: Develop Skills Online (CAN-DO) program

INTERVENTIONS:
Other: Caregiver as Navigator: Develop Skills Online (CAN-DO) program — Online, asynchronous psychoeducation program for dementia family caregivers. The program is meant to enhance caregivers' knowledge and skills for navigating healthcare, financial, legal, and family systems.
  The program has three main sections.
  * The first section provides information and how to prepare for using the healthcare system and community-based services in dementia care and support.
  * The second provides information about how to be more effective when using the financial and legal system either for yourself or your person.
  * The third section of the course provides information about ways to manage and navigate family dynamics present in various caregiving scenarios more effectively.
  Other Names: CAN-DO
Other: Healthy Living online course — Online program for dementia family caregivers about "Healthy Living" for the first 4 months post-randomization.
  Arms: Attention Control program group

SUMMARY:
This study is designed to learn more about ways to promote caregiver mastery online. 270 dementia family caregivers will be enrolled and randomized to take the CAN-DO online course immediately or after a waiting period. They will participate in interviews before and after the course; total time of study participation is 6 months.

DETAILED DESCRIPTION:
Family members and friends are the core of the uncoordinated system of care that tenuously maintains persons living with dementia in their community settings and delays their placement into more costly settings of institutional care, providing more contributed and out of pocket care support than Medicare and Medicaid combined.

The CAN-DO program fills a significant gap in caregiver psychoeducation programming by focusing not principally on day-to-day care management but on the many substantial system navigation tasks that caregivers assume. Supported by preliminary efficacy data, CAN-DO will employ state-of-the art asynchronous interactive learning methods to enhance caregivers' mastery of skills and confidence to navigate healthcare and other (legal, financial, social service, and family) systems that are crucial to the continued community living of persons affected with dementia illnesses.

This study will enroll 270 dementia family caregivers who will be randomized to take the CAN-DO course immediately or after a waiting period. They will participate in interviews before and after the course; total time of study participation is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Family member or friend providing at least 4 hours per week of informal care for a community-dwelling person living with ADRD
* 18 years or older
* Has internet access
* Does not have to co-reside with the individual
* Understands, speaks, and reads English

Exclusion Criteria:

* Family caregiver plans to move care recipient to an institutional setting within the next six months
* Care recipient currently enrolled in hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in Pearlin Caregiver Stress Scales score | Baseline, 2, 4, 6, and 8 months post-intervention
  This primary outcome will measure Caregiver Mastery (including Competence, Confidence, Management of Situation). The Pearlin caregiver scale includes 8 items, with a rating from 1-4 for each of them. Total possible score range is 8-32. Higher score correlates with better outcome.
Change in Caregiver Assessment of Behavioral Skill scale score | Baseline, 2, 4, 6, and 8 months post-intervention
  This study outcome will also measure Caregiver Mastery. Caregiver Assessment of Behavioral Skills score will be assessed using the Fortinsky scale that includes 17 items rated from 0-3 each. Possible score range is 0-51. Higher score correlates with better outcome.
Change in State-Trait Anxiety Scale score | Baseline, 2, 4, 6, and 8 months post-intervention
  This outcome will measure Caregiver Emotional Wellbeing. The State-Trait Anxiety Scale includes 20 items, each of them rated 1-4. Total possible score range 20-80 with higher score correlated with better study outcome.
Change in Perceived Stress Scale score | Baseline, 2, 4, 6, and 8 months post-intervention
  This outcome will measure Caregiver Emotional Wellbeing. The Perceived Stress Scale includes 10 items, each of them rated 1-5, with a total possible score 10-50. Lower score correlates with better study outcome.
Change in Caregiver Burden Index | Baseline, 2, 4, 6, and 8 months post-intervention
  This outcome will measure Caregiver Emotional Wellbeing. The caregiver burden Index includes 22 items, each of them rated 0-4, with a total possible score 0-88. Lower score correlates with better study outcome.
Change in Dyadic Relationship Scale score | Baseline, 2, 4, 6, and 8 months post-intervention
  This outcome will assess Caregiver Emotional Wellbeing. The Dyadic Relationship Scale includes 11 items rated from 1 to 4, with a total possible score range 11-44. Higher score correlates with better outcome.

SECONDARY OUTCOMES:
Change in Revised Memory and Behavior Problem Checklist score | Baseline, 2, 4, 6, and 8 months post-intervention
  This outcome will assess Care Recipient Quality of Life. Total possible score: 0-96; Higher score correlates with worse outcome.
Change in Quality of Life in Alzheimer's score | Baseline, 2, 4, 6, and 8 months post-intervention
  This outcome will assess Care Recipient Quality of Life. The total possible score is 13-52; Higher score correlates with better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Clevenger, RN, DNP, Principal Investigator — Emory University
Locations (1):
- Emory Roybal Center for Dementia Caregiving Mastery, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified aggregate data will be shared. Transcripts from interviews with patients and healthcare providers will be de-identified and sensitive content redacted where identification is plausible. These de-identified and redacted transcripts and coding summaries will be shared. All shared data sets and metadata will be made publicly available through Emory's Dataverse data repository. Documentation and support materials (e.g., survey questions with value sets and interview questions).
Supporting Information: ICF
Time Frame: Final data submission and release of data used in publications will occur approximately 8 and 12 months following the end of fieldwork, respectively. Datasets underlying publications will be shared at or prior to initial publication date. Data will not be published or will not be shared before the end of this award. Shared data will be preserved according to Emory's Dataverse data repository data retention policy. The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period.
Access Criteria: Data will be available by controlled access only. Research participants will receive information about where and how data from this study will be shared during study enrollment procedures and in informed consent documents. Interview participants will be informed their data will be shared on Emory's Dataverse data repository with controlled access for future use. Participants who want to withdraw their data from the study prior to de-identification may contact the study team or the university's research administration office.